CLINICAL TRIAL: NCT00351260
Title: British Bifurcation Coronary Study - Old, New and Evolving Strategies.
Brief Title: BBC ONE - British Bifurcation Coronary Study
Acronym: BBC ONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Sussex County Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COREC2006
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-03

CONDITIONS: Ischaemic Heart Diseases; Stenosis; Angina
Keywords: Bifurcation; Coronary; Stenosis; Stent; drug elution
MeSH Terms: conditions — Coronary Artery Disease; Constriction, Pathologic; Angina Pectoris | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Coronary Angioplasty

SUMMARY:
The study aims to assess whether a SIMPLE or a COMPLEX strategy is best for the treatment of coronary bifurcation stenoses.

DETAILED DESCRIPTION:
500 patients will be randomised to either a SIMPLE strategy (provisional T stenting) or a COMPLEX strategy (crush or culotte stenting) with clinical follow-up at 9 months.

ELIGIBILITY:
Inclusion Criteria:>18 years

* Coronary Bifurcation Lesion requiring treatment

Exclusion Criteria:

* Cardiogenic Shock
* Acute MI
* Additional type C lesion for Rx platelets <50
* LVEF <20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2005-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Death
Myocardial infarction
Target vessel revascularisation

SECONDARY OUTCOMES:
Repeat angiography
Stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: David J.R, Hildick-Smith, MD, Principal Investigator — Royal Sussex County Hospital
Locations (1):
- Royal Sussex County Hospital, Brighton, United Kingdom

REFERENCES:
- [Derived] Behan MW, Holm NR, de Belder AJ, Cockburn J, Erglis A, Curzen NP, Niemela M, Oldroyd KG, Kervinen K, Kumsars I, Gunnes P, Stables RH, Maeng M, Ravkilde J, Jensen JS, Christiansen EH, Cooter N, Steigen TK, Vikman S, Thuesen L, Lassen JF, Hildick-Smith D. Coronary bifurcation lesions treated with simple or complex stenting: 5-year survival from patient-level pooled analysis of the Nordic Bifurcation Study and the British Bifurcation Coronary Study. Eur Heart J. 2016 Jun 21;37(24):1923-8. doi: 10.1093/eurheartj/ehw170. Epub 2016 May 8. PMID 27161619
- [Derived] Behan MW, Holm NR, Curzen NP, Erglis A, Stables RH, de Belder AJ, Niemela M, Cooter N, Chew DP, Steigen TK, Oldroyd KG, Jensen JS, Lassen JF, Thuesen L, Hildick-Smith D. Simple or complex stenting for bifurcation coronary lesions: a patient-level pooled-analysis of the Nordic Bifurcation Study and the British Bifurcation Coronary Study. Circ Cardiovasc Interv. 2011 Feb 1;4(1):57-64. doi: 10.1161/CIRCINTERVENTIONS.110.958512. Epub 2011 Jan 4. PMID 21205942
- [Derived] Hildick-Smith D, de Belder AJ, Cooter N, Curzen NP, Clayton TC, Oldroyd KG, Bennett L, Holmberg S, Cotton JM, Glennon PE, Thomas MR, Maccarthy PA, Baumbach A, Mulvihill NT, Henderson RA, Redwood SR, Starkey IR, Stables RH. Randomized trial of simple versus complex drug-eluting stenting for bifurcation lesions: the British Bifurcation Coronary Study: old, new, and evolving strategies. Circulation. 2010 Mar 16;121(10):1235-43. doi: 10.1161/CIRCULATIONAHA.109.888297. Epub 2010 Mar 1. PMID 20194880